CLINICAL TRIAL: NCT06155838
Title: Reducing Depression and Anxiety Among Teens in Multan, Pakistan: a Cluster Randomized Controlled Trial
Brief Title: Reducing Depression and Anxiety Among Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Shandong University (Other)
Responsible Party: Principal Investigator, Lubna Ghazal, PhD student, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AgaKhanUGhazalet.al(2023)
Record Dates: First submitted 2023-04-17; First posted 2023-12-05 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Anxiety; Depression
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- EASE Intervention (Experimental): The intervention consists of four fundamental themes that have empirical support, structured across seven group sessions for adolescents and three group sessions for their parents or guardians. The sessions for teenagers will be conducted in person, spanning seven weeks with one session per week, each lasting 90 minutes. Similarly, three sessions are scheduled for parents.
  In accordance with WHO guidelines (2016), the intervention will be administered by non-specialist co-facilitators(class teachers) who possess at least 16 years of education (undergraduate degree). These co-facilitators will undergo a ten-day training program, demonstrating mock sessions as part of this training. During the intervention delivery, they will also benefit from weekly supervision provided by a specialist, who will be a graduate psychologist or trained nurse in mental health.
  Interventions: Other: "Early Adolescent Skills for Emotions (EASE)
- control/ wait list (No Intervention): Throughout the study, participants in the control group will continue to receive standard treatment. Nevertheless, following the conclusion of the trial, all control group participants will undergo the EASE intervention over a seven-week period, which will also involve three sessions for their parents and guardians. This approach ensures that the control group is not placed at a disadvantage, in alignment with ethical principles.

INTERVENTIONS:
Other: "Early Adolescent Skills for Emotions (EASE) — Weekly Schedule for Teen's and their parents Sessions:
  Over the course of 7 sessions, with one session per week lasting 90 minutes, the following core components will be covered:
  Week 1: Exploring My Feelings
  Week 2: Learning to Calm
  Week 3 & 4: Learning CBT- Restructuring My Thinking, Changing Feelings and My Actions & Managing My Emotions and Issues
  Week 5 & 6: Fostering Independent Problem-Solving Skills and Seeking Help
  Week 7: Relapse Prevention
  2.0 For parents/ guardians
  Week 3 Psychoeducation (to develop skills to be able to identify, listen, better respond and provide comfort to teens when they are overwhelmed by anxiety and depression).
  Week 4 Positive parenting strategies
  Week 5 Parents/ guardians Self-care
  Arms: EASE Intervention

SUMMARY:
The objective of this clinical trial is to assess the efficacy of the Early Adolescent Skills for Emotions (EASE) program, a school-based, non-specialist psychosocial intervention developed by the WHO for LMICs, in alleviating Anxiety and Depression among teens aged 13-19. The primary inquiries it seeks to address include:

Does the EASE intervention effectively reduce anxiety and depression scores 12 weeks after implementation?

* Can the EASE intervention enhance quality of life, improve problem-solving skills, and increase perceived emotional support?
* Is the EASE intervention beneficial for enhancing the psychological well-being of parents and fostering positive parent-teen relationships?

DETAILED DESCRIPTION:
Background:

Anxiety and depression significantly impact global adolescent mental health, with 1 in 4 adolescents requiring immediate attention. Many mental health disorders emerge in late childhood and early adolescence, worsening the burden on youth and later in life. In severe cases, suicide can occur at an alarming rate of one person every 40 seconds. In Pakistan, with a large population of 220 million, 50% aged between 12-25, the rates of anxiety and depression among adolescents are concerning. A recent study of 400 high school adolescents (15-18 years) in Pakistan revealed a prevalence of around 53% for anxiety and depression. Early preventive interventions like cognitive behaviour therapy and interpersonal therapy can empower adolescents to manage these issues, but accessing mental health services conveniently remains a challenge. Engaging mainstream academic institutions for early intervention in schools is crucial to combat anxiety, depression, and suicidal thoughts among adolescents in Pakistan.

Introduction:

Anxiety and depression pose significant psychological distress and mental health challenges for adolescents worldwide, highlighting the need for evidence-based psychological interventions tailored to teens. This study aims to assess the effectiveness of a school-based psychosocial intervention, the Early Adolescent Skills for Emotions (EASE) program developed by the WHO, in reducing psychosocial distress among adolescents aged 13-19.

Method and Analysis:

A two-parallel-arm, single-blinded, cluster randomized controlled trial will be conducted in Multan, Pakistan's school settings. Eight eligible public school clusters will be randomly allocated in a 1:1 ratio to the control arm (n=4) and intervention arm (n=4). The trial will recruit 450 adolescents (56 students from each school) experiencing psychosocial distress between April and May 2023. In the intervention arm, teens will receive the EASE program over 7 weeks, featuring psychoeducation, stress management, behavioural activation, problem-solving, and relapse prevention. Teachers will be trained in active listening, quality time spent, and the use of praise to assist their students. A qualitative study will explore facilitating and challenging factors related to intervention in low-resource school settings.

Ethical Approval:

Ethical approval has been obtained from the Ethics Committee of the School of Nursing at Shandong University, Jinan, China.

ELIGIBILITY:
Inclusion Criteria:

* Teens aged 13-19 years
* Living with parents/primary caregivers
* Enrolled in public middle and high schools of Multan, Southern Punjab, Pakistan
* Teens Assent - agreed and signed by teen
* Informed consent from parents- agreed and signed by parents

Exclusion Criteria:

* Teens part of a dysfunctional family
* Psychiatric issues
* Physical and sensory disorder diagnosis.

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 450 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Aga Khan University Anxiety and Depression Scale (AKUADS-25) | at 12 weeks' post-intervention
  AKUADS will be used to assess anxiety and depression affecting the target population. Items score ranges from 0-3 (0= never, 1=sometime, 2=mostly, 3=always) for each question item hence the total score of the tool is 0-75. The higher the score the more anxiety and depression will be severe with the cut score of 19.

SECONDARY OUTCOMES:
The Kessler Psychological Distress Scale -10 (K-10) | at 12 weeks' post-intervention
  K-10 will assess psychological distress among teens and parents. It will be measured on a scale from five to one (5=all of the time; 4= Most of the time; 3 some of the time; 2= A little of the time; 1= none of the time). The scores range from 6 to 30, by summing the individual items, total scores are calculated. The higher scores indicate high psychological distress.
The Perceived Emotional/Personal Support Scale ( PEPSS) | at 12 weeks' post- intervention
  The Perceived Emotional/Personal Support Scale ( PEPSS) measures the perceived emotional support. On a four-point scale - hardly at all 4 to very much 1. The higher scores show a lack of perceived support.
The Social Problem-Solving Inventory-Revised Short Form- 25 | at 12 weeks' post- intervention
  it measures problem-solving skills in a situation. The total score of this scale varies between 0 and 20 points. The highest scores correspond to better social problem-solving abilities.
Parent-rated Pediatric Quality of Life (PedsQL). | at 12 weeks' post- intervention
  This tool will be utilized to assess the child's quality of life (health-related). This tool measures a child's quality of health on a points Likert scale ranging from 'no problem= 1' to 'almost always a problem= 4'. "Items are then reverse-scored and linearly transformed to a 0-100 so that higher scores indicate better quality of life.
Parenting practices | at 12 weeks' post- intervention
  The assessment of parenting behaviors and practices will utilize the Alabama Parenting Questionnaire-42 (APQ-42) (Maguin, Nochajski, De Wit, & Safyer, 2016)., this tool includes five constructs : involvement (10 items), supervision and monitoring (10 items), positive parenting (6 items), consistent discipline (6 items), and corporal punishment (3 items), with the additional 7 items addressing alternative disciplinary practices. Each item, rated on a 5-point scale from 1 (never) to 5 (always), contributes to the construct's score, calculated by summing the relevant items.
The Psychological Sense of School Membership | at 12 weeks' post- intervention
  The assessment of perceived belonging and psychological engagement in school will utilize the Psychological Sense of School Membership (PSSM) scale (Goodenow, 1993). This comprehensive scale delves into the sense of belonging in school environments, focusing on caring relationships, acceptance, and rejection. Comprising 18 items rated on a likert scale from 1 (not at all true) to 5 (completely true), scores are calculated by summing responses and then averaging, resulting in a score range of 1 to 5. Higher scores signify a stronger sense of perceived belonging and engagement within the school community.
Strengths and Difficulty Questionnaire | at 12 weeks' post- intervention
  The Strengths and Difficulties Questionnaire (SDQ), a widely utilized screening tool for assessing psychological adjustment in children and adolescents (Goodman et al., 1998), categorizes positive attributes (strengths) and problematic behaviors (difficulties) across five domains, each comprising 5 items: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior (strengths). Respondents use a Likert scale ("not true= 0," "somewhat true=1," or "certainly true=2") to indicate their response, representing a three-point categorical scale. Scores within each domain are summed, with higher scores in emotional symptoms, conduct problems, hyperactivity/inattention, and peer relationship problems indicating greater difficulties, while higher scores in the prosocial behavior domain signify strengths.
Moderating Factors | T1, T2, T3
  We will also explore potential moderating factors that may influence the intervention's effectiveness on the primary outcomes. These factors include gender, age groups, socioeconomic status, parental education, and parents' psychological well-being. Statistical analyses will assess whether these variables moderate the relationship between the intervention and changes in anxiety and depression.

CONTACTS AND LOCATIONS:
Overall Officials: Lubna Ghazal, Principal Investigator — Aga Khan University; Coa Fenglin, Study Chair — Shandong University - China; Cui Naixue, Study Director — Shandong University - China
Locations (1):
- Office of the Chief Executive Officer, District Education Authority, Multan, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
As mentioned below.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: June 2026- December 2026
Access Criteria: Anyone with a reasonable reason

REFERENCES:
- [Derived] Ghazal L, Cui N, Cao F. To evaluate the EASE intervention for reducing anxiety and depression among adolescents in Pakistan: a protocol for a mixed methods study, including a cluster-randomised controlled trial. BMJ Open. 2025 Mar 22;15(3):e086393. doi: 10.1136/bmjopen-2024-086393. PMID 40122537